CLINICAL TRIAL: NCT05018091
Title: Dexamethasone in Total Knee Arthroplasty: What Dose Should we be Giving Patients Intraoperatively
Brief Title: Dexamethasone in Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Craig J Della Valle, MD, Professor of Orthopedic Surgery, Chief Division of Adult Reconstruction, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 21081102
Record Dates: First submitted 2021-08-12; First posted 2021-08-24 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Total Knee Arthroplasty
Keywords: dexamethasone; opioid consumption; postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group 1 (Active Comparator): 4mg intravenous dexamethasone, administered shortly after induction of anesthesia
  Interventions: Drug: Dexamethasone 4mg
- Group 2 (Active Comparator): 8mg intravenous dexamethasone, administered shortly after induction of anesthesia
  Interventions: Drug: Dexamethasone 8 Mg/mL Injectable Suspension
- Group 3 (Active Comparator): 16mg intravenous dexamethasone, administered shortly after induction of anesthesia
  Interventions: Drug: Dexamethasone 16mg

INTERVENTIONS:
Drug: Dexamethasone 4mg — 4mg intravenous dexamethasone, administered shortly after induction of anesthesia
  Other Names: Group 1
  Arms: Group 1
Drug: Dexamethasone 8 Mg/mL Injectable Suspension — 8mg intravenous dexamethasone, administered shortly after induction of anesthesia
  Other Names: Group 2
  Arms: Group 2
Drug: Dexamethasone 16mg — 16mg intravenous dexamethasone, administered shortly after induction of anesthesia
  Other Names: Group 3
  Arms: Group 3

SUMMARY:
The purpose of this study is to determine the most efficacious and safest dexamethasone dose given intraoperatively during total knee arthroplasty that reduces postoperative opioid consumption and pain, improves postoperative nausea and vomiting, and minimizes postoperative complications.

DETAILED DESCRIPTION:
Study design: Prospective randomized controlled trial

Scientific Background: In contemporary total joint arthroplasty (TJA), multimodal anesthesia and analgesia is used to improve postoperative pain, reduce opioid consumption, and minimize complications after surgery such as postoperative nausea and vomiting.1-3 Multiple medications with varying mechanisms of action are used at different time points throughout the perioperative period to modulate different pain receptors. Corticosteroids are a medication commonly utilized intraoperatively as part of contemporary multimodal protocols.

Corticosteroids are frequently used in TJA due to their potent anti-inflammatory and anti-emetic properties. Several studies have demonstrated that corticosteroids reduce postoperative nausea and vomiting as well as postoperative pain and opioid consumption.4-6 However, the optimal medication, dose, and number of doses of corticosteroid that should be administered in the perioperative period remain unknown. In addition, it remains unclear if corticosteroids can be safely used in patients with diabetes mellitus or if corticosteroids increase the risk of postoperative complications such as periprosthetic joint infection. Thus, the purpose of our study is to determine the most efficacious and safest dose of corticosteroids that should be administered intraoperatively during TJA.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Primary total knee arthroplasty
* Patients staying at least one night in the hospital after surgery

Exclusion Criteria:

* Same day discharge Age < 18 years Revision or partial total knee arthroplasty Corticosteroid use within 3 months prior to surgery Inflammatory arthritis Current systemic fungal infection Renal or liver failure Prior adverse reaction to corticosteroid Primary TKA requiring hardware removal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | 48-hours postoperative (after surgical intervention)
  48 hours of cumulative opioid consumption measured in oral morphine equivalents

SECONDARY OUTCOMES:
Postoperative pain scores at rest and with activity | Immediately after surgical intervention (TKA) for days 1 through 7 after surgery
  Using daily Defense and Veterans Pain Rating scale to rate pain at rest and with activity
Postoperative nausea and vomiting | Immediately after surgical intervention (TKA) for days 1 through 7 after surgery. Using numeric rating scale.
  Using numeric rating scale, (1-10, where 10 is most nausea, causing vomiting followed by number of times participant vomited in 24-hour period).
Postoperative Blood glucose levels and insulin use | Immediately following surgical intervention until discharge from hospital (up to 30 days after surgery if still in hospital)
  check glucose levels in daily blood draws when inpatient at hospital, insulin if applicable
Length of stay | immediately following surgery (intervention), number of days spent in the hospital after surgery to discharge, up to 30 days after intervention
  Days inpatient at hospital after surgery
Sleeplessness/insomnia | Immediately after surgical intervention (TKA) for days 1 through 7 after surgery, recording 24 hour sleep patterns
  recorded by patient, daily sleep schedule
Number of participants with complications (such as readmission to hospital) up to 30 days after surgical intervention | <30 days after surgical intervention, document any readmissions to the hospital or complications that occur within 30 days from the day of surgery
  Readmission after surgery, infection, VTE, GI hemorrhage or any other complication that requires rehospitalization

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Stanford University, Redwood City, California
  - University of California, San Francisco, San Francisco, California
  - Rush University medical Center, Chicago, Illinois
  - Mass General Brigham, Somerville, Massachusetts
  - Mayo Clinic Institutional Review, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - NYU Langone Health, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - University of Pennsylvania Perelman School of Medicine, Philadelphia, Pennsylvania
  - Jefferson Philadelphia University and Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moucha CS, Weiser MC, Levin EJ. Current Strategies in Anesthesia and Analgesia for Total Knee Arthroplasty. J Am Acad Orthop Surg. 2016 Feb;24(2):60-73. doi: 10.5435/JAAOS-D-14-00259. PMID 26803543
- [Background] Hannon CP, Keating TC, Lange JK, Ricciardi BF, Waddell BS, Della Valle CJ. Anesthesia and Analgesia Practices in Total Joint Arthroplasty: A Survey of the American Association of Hip and Knee Surgeons Membership. J Arthroplasty. 2019 Dec;34(12):2872-2877.e2. doi: 10.1016/j.arth.2019.06.055. Epub 2019 Jul 8. PMID 31371038
- [Background] Parvizi J, Miller AG, Gandhi K. Multimodal pain management after total joint arthroplasty. J Bone Joint Surg Am. 2011 Jun 1;93(11):1075-84. doi: 10.2106/JBJS.J.01095. PMID 21655901
- [Background] Lex JR, Edwards TC, Packer TW, Jones GG, Ravi B. Perioperative Systemic Dexamethasone Reduces Length of Stay in Total Joint Arthroplasty: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Arthroplasty. 2021 Mar;36(3):1168-1186. doi: 10.1016/j.arth.2020.10.010. Epub 2020 Oct 16. PMID 33190999
- [Background] Lunn TH, Kehlet H. Perioperative glucocorticoids in hip and knee surgery - benefit vs. harm? A review of randomized clinical trials. Acta Anaesthesiol Scand. 2013 Aug;57(7):823-34. doi: 10.1111/aas.12115. Epub 2013 Apr 15. PMID 23581549
- [Background] Chen P, Li X, Sang L, Huang J. Perioperative intravenous glucocorticoids can decrease postoperative nausea and vomiting and pain in total joint arthroplasty: A meta-analysis and trial sequence analysis. Medicine (Baltimore). 2017 Mar;96(13):e6382. doi: 10.1097/MD.0000000000006382. PMID 28353565